CLINICAL TRIAL: NCT04671290
Title: Temocillin Versus Carbapenems for Urinary Tract Infection Due to ESBL-producing Enterobacteriaceae: a Multicenter Case-control Study.
Brief Title: Temocillin Versus Carbapenems for Urinary Tract Infection Due to ESBL-producing Enterobacteriaceae
Acronym: TEMO-BLSE
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Collaborators: APHP (Other); Sorbonne University (Other); Hopitaux Civils de Colmar (Other); Hopital Foch (Other); CH Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 19-10
Record Dates: First submitted 2020-12-01; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Urinary Tract Infection Bacterial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Carbapenem (imipenem, or meropenem, or ertapenem) as first-line therapy or after receiving up to 72 hours of other antibiotics (including aminoglycosides).
  Interventions: Other: Any intervention
- Cases: Temocillin above 50% of the time of effective antibiotic therapy duration. Temocillin had to be given as first-line therapy or after receiving a maximum of 5 days of other antibiotics (including carbapenems and aminoglycosides).
  Interventions: Other: Any intervention

INTERVENTIONS:
Other: Any intervention — No intervention

SUMMARY:
To assess the efficacy of temocillin compared to carbapenems for the management of ESBL-E UTI.

DETAILED DESCRIPTION:
Adults with a definite diagnosis of ESBL-E UTI between January-2015 and October-2019 were enrolled in a multicenter retrospective case-control study. Cases were treated with temocillin ≥50% of the effective antibiotic therapy duration. Control exclusively received carbapenem over the effective antibiotic therapy duration.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Diagnosis of UTI defined by at least two of the following symptoms :chills,temperature >38°C (fever), flank or pelvic pain, nausea or vomiting, dysuria, urinary frequency, or urinary urgency, costovertebral angle tenderness on physical examination
* Positive urine culture with ≥ 103 CFU/mL of a single strain of ESBL-E
* Confirmed ESBL-producing enterobacteriaceae (ESBL-E) susceptible to carbapenems

Exclusion Criteria:

* Multibacterial infection
* Opposition to data collection according to GDPR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive adults hospitalized in participating sites for a definite diagnosis of UTI due to an ESBL-producing enterobacteriaceae (ESBL-E) susceptible to carbapenems, were eligible for the study if they provided a non-opposition form for retrospective data collection.
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
Rate of clinical cure | Day 14 (End of antibiotic treatment according to national recommendations)
  Number of patient in clinical cure is defined as the resolution of fever and symptoms of UTI present at antibiotic initiation (and no new symptoms) and the absence of clinical or microbiological failure.

SECONDARY OUTCOMES:
Kinetic of fever defervescence | Baseline (day 0), day 3, day 7, day 14
  Median fever calculation
Inflammatory biomarkers | Baseline (day 0), day 3, day 7, day 14
  White blood cells (WBC) count (/mm3)
Inflammatory biomarkers | Baseline (day 0), day 3, day 7, day 14
  CRP level (mg/l)
Length of hospital stay | 3 months after UTI diagnosis
  Mean duration of hospital stay
Relapse of UTI | 3 months after antibiotic therapy initiation
  Number of patient with a new UTI diagnosis after the end of antibiotic treatment
Loss to follow-up, re-hospitalization, and mortality (safety endpoints) | 3 months after antibiotic therapy initiation
  Number of loss to follow-up, re-hospitalization, and mortality

CONTACTS AND LOCATIONS:
Overall Officials: Mathieu LAFAURIE, M.D, Principal Investigator — APHP, St Louis Hospital

IPD SHARING:
Plan to Share IPD: No